CLINICAL TRIAL: NCT01279135
Title: Phase III Randomized Trial of Image Guided Intensity Modulated Radiotherapy (IG-IMRT) and Conventional Radiotherapy for Late Toxicity Reduction After Postoperative Radiotherapy in Ca Cervix.
Brief Title: Tomotherapy vs Conventional Radiation for Adjuvant Pelvic RT in Ca Cervix
Acronym: PARCER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Supriya Sastri (chopra), Associate Professor, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Project 803
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Cancer Cervix
Keywords: IGRT,Postoperative, Cervix, Late toxicity, Bowel
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients enrolled are randomized to either conventional arm or tomotherapy arm for treatment after stratification according to type of surgery the patient underwent and the indication of chemotherapy along with radiation
Masking Description: No masking. This is a open-label study.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional RT (Active Comparator): Patients in this arm will receive conventional radiation with or without chemotherapy
  Interventions: Radiation: Conventional Radiation
- Tomotherapy based IGRT (Experimental): Patients in this arm will receive Tomotherapy based IGRT with or without chemotherapy
  Interventions: Radiation: Tomotherapy based IGRT

INTERVENTIONS:
Radiation: Conventional Radiation — Standard Pelvic Radiation 50 Gy/ 25 fractions over 5 weeks
  Arms: Conventional RT
Radiation: Tomotherapy based IGRT — Patients in this arm will received Tomotherapy based Image Guided Intensity Modulated Radiotherapy to a dose of 50 Gy/25 fractions/5 weeks
  Arms: Tomotherapy based IGRT

SUMMARY:
The study tests Tomtherapy based Image Guided Radiation against conventional radiation techniques for it's ability to reduce long term small bowel toxicity.

DETAILED DESCRIPTION:
Postoperative pelvic radiotherapy (+/- chemotherapy) leads to reduction in the risk of local recurrence and improves progression free survival (PFS) in patients with post-operative intermediate and high risk factors following Wertheim's hysterectomy. However, adjuvant external beam radiotherapy and vaginal cuff brachytherapy increase the risk of small bowel toxicity such that patients undergoing external beam pelvic radiotherapy and vaginal cuff brachytherapy may have 15-18% incidence of late RTOG ≥ grade II small bowel toxicity. Phase II studies using new techniques like Intensity Modulated Radiotherapy (IMRT) have reported up to 50% reduction in small bowel doses with up to 30% reduction in ≥ grade II acute toxicity. However, there is no randomized data demonstrating the benefit of highly specific and conformal techniques like image guided (IG)-IMRT in reducing radiation induced small bowel toxicity in patients with cervical cancers. The present study is being proposed to test if use of IG-IMRT with Tomotherapy is associated with reduced small bowel late toxicity

ELIGIBILITY:
Inclusion Criteria:

* Histopathological diagnosis of carcinoma cervix with postoperative intermediate or high risk features.
* Age >18 years.
* Planned for Wertheim's hysterectomy or has already undergone Wertheim's hysterectomy OR has undergone Simple Hysterectomy with no evidence of residual nodes on MRI/PET imaging+/- confirmatory nodal biopsy.
* No evidence of paraaortic nodal metastasis.

Exclusion Criteria:

* History of multiple previous abdominal surgeries placing patient at baseline high risk of bowel toxicity or any other medical condition with baseline bowel movement disorder.
* Rectal Polyps or extensive hemorrhoids.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Late bowel toxicity ≥ Grade II | Median follow up of 3 years
  Time to event and severity of late bowel toxicity are assessed

SECONDARY OUTCOMES:
To identify small bowel dose volume characteristics that predict for ≥ Grade II late toxicity | Median follow up of 3 years
  Data on dosimetric analysis of small bowel dose in reference to volume are collected in both arms and assessed for predicting dose prescription for ≥ grade II late bowel toxcity
To evaluate acute toxicity difference in two study arms using CTCAE version 3.0 | Within 90 days
  Acute toxicity will be reported using CTCAE V.3.0. CTCAE forms will be filled before starting radiation, weekly during radiation treatment and on each scheduled follow-up. If any toxicity occurs at another time point additional forms will be filled to capture the same. Acute toxicity difference will be calculated between the two study arms.
Preoperative functional imaging features that predict for local and distant recurrence will be identified | 3 years after completion of accrual
  Images acquired pre-operatively are analysed for features that predict local and distant recurrence.
To compare quality of life between Tomotherapy vs conventional radiotherapy arm using EORTC QLQ C30 | 3 years from completion of accrual
  Assessment is done for all enrolled patients to compare the quality of life after treatment with tomotherapy and conventional radiation . EORTC QLQC30 module will be used for evaluating QOL of patients. QOL scoring will be done as per standard recommendations outlined in EORTC QLQ C30 scoring manual. All patients will undergo QOL evaluation at baseline, after treatment and at subsequent follow-up. Scale- Not at all-1 , A little Bit-2, Quite a bit-3, very much-4.
  1 will be considered as better outcome & 4 will be considered as worst outcome.
To compare quality of life between Tomotherapy vs conventional radiotherapy arm using EORTC QLQ CX24 | 3 years from completion of accrual
  Assessment is done for all enrolled patients to compare the quality of life after treatment with tomotherapy and conventional radiation. EORTC QLQCX24 module will be used to assess disease-specific and treatment-specific aspects of QoL in patients with cervical cancer. CX24 QOL scoring will be done as per standard recommendations outlined in EORTC QLQ CX24 scoring manual. All patients will undergo QOL evaluation at baseline, after treatment and at subsequent follow-up.
  Scale- Not at all-1 , A little Bit-2, Quite a bit-3, very much-4.
  1 will be considered as better outcome & 4 will be considered as worst outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Supriya Chopra, MD,DNB, Principal Investigator — ACTREC, Tata Memorial Centre
Locations (1):
- Advanced Centre for Treatment, Research and Education in Cancer, Tata Memorial Centre, Navi Mumbai, Maharashtra, India

REFERENCES:
- [Background] Chopra S, Engineer R, Mahantshetty U, Misra S, Phurailatpam R, Paul SN, Kannan S, Kerkar R, Maheshwari A, Shylasree Ts, Ghosh J, Gupta S, Thomas B, Singh S, Sharma S, Chilikuri S, Shrivastava SK. Protocol for a phase III randomised trial of image-guided intensity modulated radiotherapy (IG-IMRT) and conventional radiotherapy for late small bowel toxicity reduction after postoperative adjuvant radiation in Ca cervix. BMJ Open. 2012 Dec 12;2(6):e001896. doi: 10.1136/bmjopen-2012-001896. Print 2012. PMID 23242243
- [Derived] Supriya C, Nilesh R, Mayuri C, Sadhana K, Reena E, Tapas D, Lavanya G, Prachi M, Amita M, Shylasree TS, Shyam S, Sudeep G. Late toxicity within a Phase III clinical trial of IG-IMRT in cervix cancer (PARCER): Reanalysis with time weighted adverse event reporting (MOSES). Radiother Oncol. 2022 Dec;177:16-20. doi: 10.1016/j.radonc.2022.10.013. Epub 2022 Oct 18. PMID 36270474
- [Derived] Chinnachamy AN, Chopra S, Krishnatry R, Kannan S, Thomas B, Mahantshetty U, Engineer R, Shrivastava SK. Evaluation of interobserver and interscale agreement in assessing late bowel toxicity after pelvic radiation in patients with carcinoma of the cervix. Jpn J Clin Oncol. 2013 May;43(5):508-14. doi: 10.1093/jjco/hyt028. Epub 2013 Mar 20. PMID 23515269